CLINICAL TRIAL: NCT03039595
Title: An Observational Study to Correlate the Results of Ploidy and Stroma Analysis With Prognosis in Early Rectal Cancer
Brief Title: Ploidy and Stroma in Early Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Chris Cunningham, Consultant colorectal surgeon, Oxford University Hospitals NHS Trust
Other Study IDs: 11846
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-03

CONDITIONS: Rectal Cancer
Keywords: Early rectal cancer; Ploidy; Tumour:stroma ratio
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ploidies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Specimens of early rectal cancer removed by transanal endoscopic microsurgery, which are routinely retained, will be further analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ploidy and tumour:stromal ratio measurements — Ploidy and tumour:stromal ratio measurements will be made on specimens of early rectal cancer removed by transanal endoscopic microsurgery (TEM)

SUMMARY:
Early rectal cancer can be removed by minimally-invasive surgery, and the standard pathological assessment of the removed tumour gives valuable information about how advanced the tumour is. This gives an indication of how likely the cancer is to recur, so doctors and patient can decide on the most appropriate further treatment and follow-up. However there is still much uncertainty in these predictions about recurrence. This study will assess two further pathology tests, ploidy and stroma ratio in the tumour, by correlating the results with outcome. This will determine whether these two tests provide additional value in predicting outcome. If so, clinicians would be better able to advise patients with early rectal cancer about their prognosis and further management.

DETAILED DESCRIPTION:
Early rectal cancer can be removed by minimally-invasive surgery, and the standard pathological assessment of the removed tumour gives valuable information about how advanced the tumour is. This information is very important in indicating whether the cancer is likely to recur, and therefore in advising the patient after surgery whether further treatment is advisable, and if not, what is the most appropriate follow-up regime. However there is still a lot of uncertainty in these predictions about recurrence of the cancer, and better tests are being sought. This study aims to look at two further pathology tests, ploidy and stroma ratio in the tumour, and correlate these test results with outcome in patients who have had an early rectal cancer removed. This will allow the investigators to assess whether these two tests provide additional value in predicting outcome. If so, clinicians would be better able to advise patients with early rectal cancer about their prognosis and further management.

Routine histopathology analysis of a rectal cancer specimen removed at surgery includes assessment of tumour size, depth of invasion, vascular, lymphatic and perineural invasion, tumour involvement of resection margins and nodal involvement. This information is valuable in predicting outcome. For example, predicted rates of local recurrence at 36 months following local excision of rectal cancer by transanal endoscopic microsurgery (TEM) based on tumour size, depth of invasion and lymphatic invasion have been tabulated. However such models are not perfect, and leave room for improvement. Ploidy and stroma ratio are two further tests which have shown some promise in predicting outcome.

Ploidy refers to the number of sets of chromosomes in a cell nucleus. Most human cells are normally diploid, with two sets of 23 chromosomes. Abnormal tumour cells may have a different number of sets of chromosomes, or be aneuploid, having some replicated or deleted chromosomes. In general, aneuploidy in cancer cells is associated with a worse prognosis. An early study of DNA ploidy in rectal cancer using flow cytometry showed an independent but small predictive effective of aneuploidy on survival. Technological advances now allow more accurate and detailed assessment of ploidy. The DNA ploidy status of tumour cells in early ovarian cancer has been found to predict which patients will benefit from adjuvant chemotherapy after surgery to remove the ovarian tumour and is used routinely in some centres to aid in decision-making.

Stroma ratio refers to the tumour: stroma ratio. A lower proportion of tumour cells or, conversely, a higher percentage of stroma, in a cancer tends to be associated with a poorer prognosis. This ratio has been found to be strongly associated with tumour growth and invasion in colorectal cancers, and to independently predict survival in patients undergoing surgery to removal colorectal tumours. However previous studies have looked mainly at more advanced colon cancers, rather than early rectal cancers, and have used only cancer-related death as the endpoint, rather than looking at local recurrence and response to adjuvant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent (in English) for participation in the study, or gave informed consent for donation of tissue for research at the time of surgery
* Male or Female, aged 18 years or above
* Diagnosed with operable rectal cancer
* Due to undergo, or has already undergone, TEM surgery to remove rectal cancer
* A useable tissue sample has already been, or will be, taken as part of routine surgery

Exclusion Criteria:

* Age less than 18
* Adults who are not able to give consent or who are deemed vulnerable
* Participants who do not have a useable tissue sample will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with rectal cancer that is operable and patients who have already had rectal cancer removed by transanal endoscopic microsurgery (TEM) in Oxford since 2007.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cunningham, MD, Principal Investigator — Employee
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual data will be made available

REFERENCES:
- [Background] Bach SP, Hill J, Monson JR, Simson JN, Lane L, Merrie A, Warren B, Mortensen NJ; Association of Coloproctology of Great Britain and Ireland Transanal Endoscopic Microsurgery (TEM) Collaboration. A predictive model for local recurrence after transanal endoscopic microsurgery for rectal cancer. Br J Surg. 2009 Mar;96(3):280-90. doi: 10.1002/bjs.6456. PMID 19224520
- [Background] Goh HS, Jass JR, Atkin WS, Cuzick J, Northover JM. Value of flow cytometric determination of ploidy as a guide to prognosis in operable rectal cancer: a multivariate analysis. Int J Colorectal Dis. 1987 Feb;2(1):17-21. doi: 10.1007/BF01648992. PMID 3598327
- [Background] Kristensen GB, Kildal W, Abeler VM, Kaern J, Vergote I, Trope CG, Danielsen HE. Large-scale genomic instability predicts long-term outcome for women with invasive stage I ovarian cancer. Ann Oncol. 2003 Oct;14(10):1494-500. doi: 10.1093/annonc/mdg403. PMID 14504048
- [Background] Park JH, Richards CH, McMillan DC, Horgan PG, Roxburgh CSD. The relationship between tumour stroma percentage, the tumour microenvironment and survival in patients with primary operable colorectal cancer. Ann Oncol. 2014 Mar;25(3):644-651. doi: 10.1093/annonc/mdt593. Epub 2014 Jan 23. PMID 24458470
- [Background] Downey CL, Simpkins SA, White J, Holliday DL, Jones JL, Jordan LB, Kulka J, Pollock S, Rajan SS, Thygesen HH, Hanby AM, Speirs V. The prognostic significance of tumour-stroma ratio in oestrogen receptor-positive breast cancer. Br J Cancer. 2014 Apr 2;110(7):1744-7. doi: 10.1038/bjc.2014.69. Epub 2014 Feb 18. PMID 24548861
- [Background] West NP, Dattani M, McShane P, Hutchins G, Grabsch J, Mueller W, Treanor D, Quirke P, Grabsch H. The proportion of tumour cells is an independent predictor for survival in colorectal cancer patients. Br J Cancer. 2010 May 11;102(10):1519-23. doi: 10.1038/sj.bjc.6605674. Epub 2010 Apr 20. PMID 20407439

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients: All patients. This is an observational study; no interventions were used.
Period: Overall Study
Arm/Group | Patients
Started | 150
Completed | 143
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Patients: All patients
Arm/Group | Patients
Number analyzed (Participants) | 143
Age, Continuous [Median (Full Range); unit: years] | 69 [38 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 143
Tumour stage [Count of Participants; unit: Participants] — Tumour component of the TNM (Tumour, Node, Metastasis) staging system determined by histopathological analysis of the resected tumour.
  Participants
    pT1 (tumour confined to the inner layer of the bowel) | 76
    pT2 (tumour extends into the muscle layer of the bowel wall) | 58
    pT3 (tumour has reached the outer lining of the bowel wall) | 9
Post-TEM management [Count of Participants; unit: Participants]
  Surveillance | 88
  Completion radical surgery | 13
  Adjuvant radiotherapy | 42

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Ploidy Status With Local Recurrence of Cancer
Description: Results of ploidy status will be correlated with patient follow-up information for between 6 months and 9 years following surgery, to look for any correlation with local recurrence of the rectal cancer
Time Frame: a minimum of 6 months after surgery
Population: Only patients for whom ploidy status was available were included in the analysis (ploidy assessment failed in 3 patients for technical reasons)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 140
Participants
  Diploid - Local recurrence | 3
  Diploid - No local recurrence | 31
  Non-diploid - Local recurrence | 14
  Non-diploid - No local recurrence | 92

2. Primary Outcome: Correlation Between Tumour: Stroma Ratio With Local Recurrence of Cancer
Description: Results of tumour:stromal ratio (TSR) will be correlated with patient follow-up information for between 6 months and 9 years following surgery, to look for any correlation with local recurrence of the rectal cancer. A 50% cut-off is used to define high TSR.
Time Frame: a minimum of 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 143
Participants
  High TSR - Local recurrence | 2
  High TSR - No local recurrence | 9
  Low TSR - Local recurrence | 17
  Low TSR - No local recurrence | 115

3. Secondary Outcome: Correlation Between Ploidy Status and Overall Survival After TEM Surgery to Remove Rectal Cancer
Description: Results of ploidy status will be correlated with patient follow-up information for between 6 months and 9 years following surgery, to look for any correlation between the test results and overall survival
Time Frame: a minimum of 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 140
Participants
  Diploid - Alive | 27
  Diploid - Deceased | 7
  Non-diploid - Alive | 86
  Non-diploid - Deceased | 20

4. Secondary Outcome: Correlation Between Tumour:Stroma Ratio and Overall Survival After TEM Surgery to Remove Rectal Cancer
Description: Results of tumour:stromal ratio (TSR) will be correlated with patient follow-up information for between 6 months and 9 years following surgery, to look for any correlation between the test results and overall survival. High TSR is defined using a 50% cut-off.
Time Frame: a minimum of 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 143
Participants
  High TSR - Alive | 6
  High TSR - Deceased | 5
  Low TSR - Alive | 110
  Low TSR - Deceased | 22

ADVERSE EVENTS:
Time Frame: Up to 12 years following surgery
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 27/143
Serious Adverse Events (participants affected / at risk) | 0/143
Other Adverse Events (participants affected / at risk) | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT03039595/Prot_SAP_000.pdf